CLINICAL TRIAL: NCT07059455
Title: Comparıson Of Analgesıc Effectıveness Of Erector Spınae Plane Block and Transmuscular Quadratus Lumborum Block In Kıdney Transplantatıon
Brief Title: Erector Spınae Plane Block and Transmuscular Quadratus Lumborum Block In Kıdney Transplantatıon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Tahsin Şimşek, ASSOCİATED PROFESSOR, Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2015/514/154/11
Record Dates: First submitted 2025-06-23; First posted 2025-07-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-06

CONDITIONS: Kidney Transplant
Keywords: erectör spiane block; Quadratus lumborum block
MeSH Terms: interventions — Parapsychology; Dental Occlusion; Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- erectör spinae plane block (Active Comparator): Erector spinae plane block (ESPB) is a regional fascial plane block method developed in recent years. In this method, analgesia is provided by injecting local anesthetic between the transverse process and the erector spinae muscles and anesthetizing the dorsal and ventral branches of the regional spinal nerves. It has a wide range of use in thoracic, lumbar, and thoracic and abdominal surgeries
  Interventions: Other: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®)
- Transmuskuler quadratus lumborum block (Active Comparator): Transmuscular quadratus lumborum block (TMQLB) is a nerve block technique in which local anesthetic is applied to the fascial plane between the psoas major (PM) and quadratus lumborum (QL) muscles. Anatomical evidence has shown that local anesthetic can spread through the thoracolumbar fascia into the thoracic paravertebral space, thus infiltrating the thoracic spinal nerves and sympathetic trunk, providing both somatic and visceral analgesia for abdominal surgery
  Interventions: Other: Quadratus Lumborum (QL) Block

INTERVENTIONS:
Other: Erector Spinae (ESP) Block with Bupivacaine (Marcaine®) — Under general anesthesia, patients in the ESP group will be positioned in the left or right lateral decubitus position, depending on the side of the surgical procedure. After the T10 spinous process is identified by manual examination, sterile conditions will be established. The transverse process and erector spinae muscles will be visualized using an ultrasound probe. Using an in-plane technique, 20 ml of 0.25% bupivacaine will be injected between the transverse process and erector spinae muscles using a 22-gauge blocking needle.
  Arms: erectör spinae plane block
Other: Quadratus Lumborum (QL) Block — Following standard anesthesia monitoring, patients will be placed in the lateral decubitus position. After the field is sterilized, a 2-5 MHz convex ultrasound probe (Samsung, HM70 EVO) will be placed between the iliac crest and costal arch at the level of the posterior axillary line. The transverse process of the L4 vertebra, erector spinae, QL, and PM muscles will be visualized. After inducing local anesthesia with 2% lidocaine (2 ml), a blocking needle (22G*100 mm, Braun) will be advanced from posterolateral to anteromedial, inserting it between the QL and PM muscles, and 20 ml of 0.25% bupivacaine will be injected.
  Arms: Transmuskuler quadratus lumborum block

SUMMARY:
Perioperative anesthesia and pain management are among the difficult situations for anesthesiologists to manage in kidney transplant patients. These patients are often complicated by comorbidities related to chronic kidney disease. The main issues in postoperative pain management for kidney transplant patients include dose adjustment, prevention of further renal damage, and maintenance of graft perfusion. Pain management in patients with end-stage renal disease may be inadequate due to limited options of systemic analgesics. In addition, regional analgesia techniques can be considered to avoid the adverse effects of anesthetics and systemic analgesics (1).

Erector spinae plane block (ESPB) is a regional fascial plane block method developed in recent years. In this method, analgesia is provided by injecting local anesthetic between the transverse process and the erector spinae muscles and anesthetizing the dorsal and ventral branches of the regional spinal nerves. It has a wide range of applications including thoracic, lumbar, and thoracic and abdominal surgeries (2,3).

Transmuscular quadratus lumborum block (TMQLB) is a nerve block technique in which local anesthetic is applied to the fascial plane between the psoas major (PM) and quadratus lumborum (QL) muscles. Anatomical evidence has shown that local anesthetic can spread through the thoracolumbar fascia into the thoracic paravertebral space, thus infiltrating the thoracic spinal nerves and sympathetic trunk, providing both somatic and visceral analgesia for abdominal surgery (4).

This study aims to evaluate the analgesic efficacy of ESPB and TMQLB in terms of pain management after kidney transplantation. The primary aim of the study was to evaluate pain scores and analgesic consumption between groups in the 24-hour postoperative period. The secondary aim was to evaluate the time to first analgesic requirement after block, the number of patients requiring analgesics, and the levels of nausea and vomiting.

DETAILED DESCRIPTION:
MATERIAL AND METHODS A total of 50 patients are planned to be included in this single-blind, prospective randomized controlled study planned to be conducted between June 10, 2025 and October 10, 2025 in the general surgery operating room of Kartal Dr. Lütfi Kırdar City Hospital.

All patients taken to the operating room will be subjected to standard monitoring techniques including temperature monitoring, electrocardiography (ECG), peripheral oxygen saturation (SpO2), end tidal carbon dioxide monitoring (EtCO2) and non-invasive blood pressure measurement, and then one of two regional anesthesia methods will be applied to the patients. Then, the surgical procedure will be started after standard general anesthesia induction and endotracheal intubation will be applied to the patients. 100 mg tramadol and 1 gr paracetamol will be administered to all patients iv for analgesia 15 minutes before the end of the operation, and 10 mg metoclopramide will be administered to patients iv for nausea and vomiting.

Randomization Patients will be divided into two groups as Group TMQLB; n=25 and Group ESPB; n=25 in a system where random numbers generated by the computer (SPSS v23.0, IBM, NewYork, USA) are used, with a ratio of 1:1. The physician who will follow up the patients postoperatively will be blind to the groups.

Power analysis As a result of the power analysis conducted for our study; the standard effect size was determined as 0.72 with a 5% margin of error and 80% power. It was decided to include a total of 50 cases, n=25 cases in each group.

Block application After regional sterile conditions are provided with 10% povidone iodine solution while the patient is in the supine position, 6-13 Mhz linear ultrasonography (USG Esaote, Via E. Melen, 77 16152 Genova, Italy) will be used for imaging for ESPB, 22 G and 100 mm block needle (Stimuplex® Ultra 360® B-Braun medical, Melsungen, Germany) will be inserted between the transverse process and the erector spinae muscle at the level of the T10 vertebra and 30 ml of a local anesthetic solution consisting of 0.25% bupivacaine will be administered to the side to be treated.

For imaging for TMQLB, 2-5 Mhz convex ultrasonography (USG Esaote, Via E. Melen, 77 16152 Genova, Italy) will be used, the transverse process will be visualized at the level of the L3 vertebra with a 22 G and 100 mm block needle (Stimuplex® Ultra 360® B-Braun medical, Melsungen, Germany), and 30 ml of a local anesthetic solution consisting of 0.25% bupivacaine will be administered to the side to be treated.

Standard postoperative analgesia protocol

1 g paracetamol will be administered intravenously to all patients every 8 hours during the postoperative 24-hour period. If the visual analog scale (VAS) values of the patients were 4 and above during follow-up, tramadol 100 mg was administered as an intravenous rescue analgesic.

Postoperative pain assessment Patients' pain levels will be assessed using a 10-point VAS at 0, 1, 2, 6, 12, and 24 hours. No pain will be assessed as 0 points, and severe pain will be assessed as 10 points. VAS scores, time to first analgesic requirement, and total tramadol consumption will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplantation
* Patients between the ages of 18-65

Exclusion Criteria:

* Patients who do not agree to participate in the study,
* Patients havecoagulopathy, liver function problems, local anesthetic allergy
* Body mass index (BMI) > 40

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
evaluate pain scores and analgesic consumption between groups | postoperative 24 hours
  Patients' pain levels will be measured at 0, 1, 2, 6, 12, and 24 hours using a 10-point VAS. No pain will be assessed as 0 points, and severe pain will be assessed as 10 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Kartal Dr Lutfi Kirdar City Hospital, Istanbul, Kartal, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided